CLINICAL TRIAL: NCT05375357
Title: Evaluation of Healing Time and Postoperative Morbidity After Implant Uncovering With Vestibularly Repositioned Flap Associated With Leucocyte Platelet Rich Fibrin (L-PRF): a Randomized and Controlled Clinical Trial
Brief Title: Platelet Rich Fibrin in Soft Tissue Healing After Implant Uncovering
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Michele Paolantonio, Full time professor, G. d'Annunzio University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19102021
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-05

CONDITIONS: Healing Surgical Wounds
Keywords: Platelet Rich Fibrin; Wound Healing; Implant Uncovering

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APF + L-PRF (Experimental): Application of a layer of L-PRF to protect the donor area after uncovering implant procedure using Apically Positioned Flap (APF).
  Interventions: Procedure: Application of L-PRF on the donor area
- APF without L-PRF (Active Comparator): The donor area is left to heal by secondary intention after APF in the implant uncovering procedure.
  Interventions: Procedure: Secondary intention healing of the donor area

INTERVENTIONS:
Procedure: Application of L-PRF on the donor area — After implant uncovering procedure with apically positioned flap, the donor area is covered with a layer of L-PRF
  Arms: APF + L-PRF
Procedure: Secondary intention healing of the donor area — After implant uncovering procedure with apically positioned flap, the donor area is left to heal by secondary intention
  Arms: APF without L-PRF

SUMMARY:
This study represents a prospective, controlled and randomized clinical trial assessing the effects of L-PRF on the healing time of the donor area and on the patient's postoperative morbidity in the 4 weeks following the Apically Positioned Flap (APF) procedure in the uncovering phase of two-stage implants.

A total of 40 patients were recruited and divided into two groups. The implant uncovering procedure in the test group was performed with APF and application of L-PRF on the donor area. Patients in the control group, on the other hand, were treated with APF alone, leaving the donor area to heal by secondary intention.

ELIGIBILITY:
Inclusion Criteria:

* to have at least one implant in the maxilla with a quantity of vestibular keratinized gingiva < 2 mm
* to be in good systemic health
* to have a good oral hygiene (FMPS and FMBS < 20%)

Exclusion Criteria:

* systemic diseases: coagulation disorders; medications affecting periodontal status in the previous 6 months; pregnancy or lactation;
* smoking habits;
* peri-implant surgery on the experimental sites.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Complete re-epithelialization of the wound of donor area (CWE) | 4 weeks
  Time needed to obtain a complete re-epithelialization of the wound of donor area

SECONDARY OUTCOMES:
Post-Operative Discomfort (D) | 4 weeks
  Evaluation of post-operative discomfort using Visual Analogue Scale (VAS).The scale is represented by a straight horizontal line of fixed length, generally 10 cm. Extremities are defined as extreme limits of the parameter to be measured, oriented from left (worst) to right (best).
Changes in Feedind Habits (CFH) | 4 weeks
  Evaluation of changes in patients' feedind habits using Visual Analogue Scale (VAS).The scale is represented by a straight horizontal line of fixed length, generally 10 cm. Extremities are defined as extreme limits of the parameter to be measured, oriented from left (worst) to right (best).
Consumption of Analgesics (AU) | 4 weeks
  Assessment of postoperative pain by the number of analgesics taken
Alteration of Sensivity (AS) | 4 weeks
  Evaluation of alteration of sensivity on donor area

CONTACTS AND LOCATIONS:
Locations (1):
- G. D'Annunzio University, Chieti, Italy

IPD SHARING:
Plan to Share IPD: No